CLINICAL TRIAL: NCT01982890
Title: Telomere Shortening as a Prognostic Marker in Early Inflammatory Arthritis: Establishing the Stability of Telomeres in Normal Individuals
Brief Title: Telomeres and T-cell Receptor Excision Circles (TRECs) From Peripheral Blood in Normal Subjects Over Time
Status: Enrolling by invitation | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Gilles Boire, Doctor, Université de Sherbrooke
Other Study IDs: Telomeres and TREC
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Telomere Length in Healthy Controls
Keywords: Telomere length; Longitudinal observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Genomic DNA extracted from peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal human controls: Observational study. Subjects are screened for the absence of severe illnesses and followed prospectively with sequential blood draws, noting the occurence of acute and chronic severe illnesses.
  Subjects are matched by age groups and sex with patients of the prospective cohort EUPA including patients with recent-onset inflammatory polyarthritis.
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — No intervention as this group is simply followed prospectively.

SUMMARY:
The Investigators have established a cohort of patients with recent-onset inflammatory arthritis called Early Undifferentiated PolyArthritis (EUPA). This cohort was established to define novel biomarkers of poor outcomes. We want to study telomere length and T-cell Receptor Excision Circles (TREC) numbers in peripheral blood as new biomarkers.

This cohort of normal controls was established to be able to define the stability over short periods of time of telomere length and TREC numbers in normal individuals, in order to compare with arthritis patients.

DETAILED DESCRIPTION:
It is difficult to establish early on the prognosis of patients with recent-onset polyarthritis. We want to know if we can use the length of telomeres in peripheral blood cells at baseline as a novel prognostic marker.

In order to be able to interpret our observations in arthritis patients over time, we need to compare these results with those observed in normal human controls adjusted for gender and for age groups.

These patients are first screened for the presence of acute or chronic severe diseases (cancer, cardiovascular, articular, et...). They then have genomic DNA extracted from peripheral blood at Baseline and at 3 months interval for a year than annually for a total duration of 5 years. A complete blood count is collected at each blood draw. At each blood draw, the appearance of acute or chronic diseases is noted.

ELIGIBILITY:
Inclusion Criteria:

Healthy-for-age subjects, as defined by Absence of acute infectious, traumatic or immunologic disease; Absence of severe chronic diseases Age and sex concordant with the stratification of patients from a longitudinal cohort of early inflammatory arthritis (EUPA)

Exclusion Criteria:

History of cancer (except a single episode of non-melanocytic skin cancer) Severe cardiovascular disease (i.e. difficult to control or requiring multiple drugs) Chronic infection Inflammatory arthritis Severe high blood pressure or diabetes (i.e. difficult to control or requiring multiple drugs) Any severe disease affecting function or difficult to control or requiring multiple drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal human controls apparied for gender and for groups of age with patients of the EUPA cohort (with inflammatory arthritis of between 1 and 12 months duration presenting for clinical care at the Rheumatology Division of the Centre hospitalier universitaire de Sherbrooke.)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-01-04 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of variability of multiple measures of the length of telomeres over one year | Over one year
  Blood draws to collect genomic DNA both from total peripheral blood cells and from peripheral blood mononuclear cells are done at 0, 3, 6, 9 and 12 months (along with a complete blood count). At each time, patients are assessed for severe acute and chronic diseases

SECONDARY OUTCOMES:
TREC numbers in peripheral blood over time | At 3, 6, 9, 12, 18, 24, 36, 48 and 60 months
  Blood draws at these time points. T cell Excision Circles are measured from genomic DNA at the same time as is telomere length
Estimation of the variability of the measure of length of telomeres with multiple measures over 5 years | 5 years
  From the end of the first year, patients will be followed yearly with an assessment of the occurence of new severe acute and chronic diseases and a blood draw to collect genomic DNA isolated from total blood cells and from isolated blood mononuclear cells, along with a complete blood count to assess lymphocyte numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boire, MD, MSc, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada